CLINICAL TRIAL: NCT05673460
Title: A Phase 1 Clinical Study of Nemtabrutinib (MK-1026) in Japanese Participants With Hematological Malignancies (BELLWAVE-002)
Brief Title: A Clinical Study of Nemtabrutinib in Japanese Participants With Hematological Malignancies (MK-1026-002)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1026-002; MK-1026-002 (Other: MSD); jRCT2031220583 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-01-04; First posted 2023-01-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Mature B-cell Neoplasms
MeSH Terms: interventions — ARQ531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nemtabrutinib (Experimental): Participants receive nemtabrutinib at specified dose orally once daily (QD) until progressive disease (PD) or discontinuation
  Interventions: Drug: Nemtabrutinib

INTERVENTIONS:
Drug: Nemtabrutinib — Nemtabrutinib tablets will be administered orally QD at dosage of 45 mg or 65 mg
  Other Names: MK-1026; ARQ 531

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of nemtabrutinib in Japanese participants with mature B-cell neoplasms.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Histologically confirmed B-cell malignancy:

  * Chronic lymphocytic leukemia (CLL)
  * Small lymphocytic lymphoma (SLL)
  * Waldenström's macroglobulinemia (WM),
  * Lymphoplasmacytic lymphoma (LPL)
  * Other B-cell neoplasm
* Failed or intolerant to either at least 2 prior regimens given in combination or sequentially OR have received 1 prior Bruton's tyrosine kinase (BTK)-containing regimen when a BTK inhibitor is approved as first line therapy
* Have the ability to swallow and retain oral medication
* Is Japanese

Exclusion Criteria:

* Active Hepatitis B virus (HBV)/Hepatitis C virus (HCV) infection at study entry
* History of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 3 years
* Known history of human immunodeficiency virus (HIV) infection
* Clinically significant gastrointestinal abnormalities that might alter absorption (eg, gastric bypass surgery, gastrectomy)
* Underlying history of severe bleeding disorders
* History or concurrent condition of pneumonitis/interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants who Experience Dose Limiting Toxicities (DLTs) per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 | Up to approximately 4 weeks
  A DLT consists of one or more of the following toxicities: Grade ≥3 nonhematologic toxicity with exception of Grade 3 nausea, vomiting, diarrhea, rash, fatigue, and uncontrolled hypertension; Grade 4 hematologic toxicity lasting >7 days, Grade 4 platelet count decreased of any duration (with exceptions), or Grade 3 platelet count decreased with bleeding, or Grade 3 or higher febrile neutropenia of any duration; Grade 3 or Grade 4 nonhematologic laboratory abnormality, if values result in drug induced liver injury (DILI), or medical intervention is required, or the abnormality leads to hospitalization, or the abnormality persists for >1 week (with exceptions); missing >25% of nemtabrutinib doses as a result of drug-related AE(s); Grade 5 toxicity. Toxicities will be graded using NCI-CTCAE version 5.0 except hematologic toxicities in participants with chronic lymphocytic leukemia (CLL) assessed according to the International Workshop on CLL (iwCLL) criteria.
Number of Participants who Experience Adverse Events (AEs) | Up to approximately 38 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Discontinuing Study Treatment due to AEs | Up to approximately 38 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Area under the Curve (AUC) of Nemtabrutinib | Day 1 of Cycles 1 and 2: Pre-dose,1, 2, 4, 6, 8, 10, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2 and 4 hours post-dose (up to ~57 days). Each cycle is 28 days
  AUC is the area under the curve of plasma concentration of nemtabrutinib. Blood samples collected at designated timepoints will be used to determine AUC.
Maximum Concentration (Cmax) of Nemtabrutinib | Day 1 of Cycles 1 and 2: Pre-dose,1, 2, 4, 6, 8, 10, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2 and 4 hours post-dose (up to ~57 days). Each cycle is 28 days
  Cmax is the maximum concentration of nemtabrutinib observed in plasma. Blood samples collected at designated timepoints will be used to determine Cmax.
Time to Maximum Concentration (Tmax) of Nemtabrutinib | Day 1 of Cycles 1 and 2: Pre-dose,1, 2, 4, 6, 8, 10, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2 and 4 hours post-dose (up to ~57 days). Each cycle is 28 days
  Tmax is the time to reach maximum concentration of nemtabrutinib. Blood samples collected at designated timepoints will be used to determine Tmax.
Minimum Concentration (Cmin) of Nemtabrutinib | Day 1 of Cycles 1 and 2: Pre-dose, 1, 2, 4, 6, 8, 10, and 24 hours post-dose; Day 1 of Cycle 3: pre-dose and 2 and 4 hours post-dose (up to ~57 days). Each cycle is 28 days
  Cmin is the minimum concentration of nemtabrutinib observed in plasma. Blood samples collected at designated timepoints will be used to determine Cmin.
Objective Response Rate (ORR) as Assessed by Investigator | Up to approximately 38 months
  ORR is the proportion of participants in the analysis population with objective response. Objective response is defined as participants who achieve at least a partial response (PR) per disease-specific criteria as assessed by investigator.
Duration of Response (DOR) as Assessed by Investigator | Up to approximately 38 months
  For participants who demonstrate an objective response as assessed by investigator, per disease-specific criteria, duration of response is defined as the time from the first documented evidence of an objective response until disease progression or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (7):
- Japan (7):
  - Nagoya University Hospital ( Site 0003), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 0002), Kashiwa, Chiba
  - Kindai University Hospital ( Site 0006), Sayama, Osaka
  - Chiba Cancer Center ( Site 0005), Chiba
  - Kyushu University Hospital ( Site 0008), Fukuoka
  - Okayama University Hospital ( Site 0007), Okayama
  - Yamagata University Hospital ( Site 0001), Yamagata

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/